CLINICAL TRIAL: NCT07386457
Title: Dimensional Changes During Early Healing Following Subepithelial Connective Tissue Graft for Root Coverage
Brief Title: Taking Measurements of a Gum Graft Site as it Heals
Status: Not yet recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Binnaz Leblebicioglu, Professor, Ohio State University
Other Study IDs: 2025H0007
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Grafting Surgery Recipients: Patients at the Graduate Periodontics Clinic at The Ohio State University who are having a gingival graft done to treat gingival recesssion.
  Interventions: Procedure: Gingival graft surgery to treat gingival recession

INTERVENTIONS:
Procedure: Gingival graft surgery to treat gingival recession — Subepithelial connective tissue grafting (SCTG) is a common procedure for the treatment of gingival recession and involves the autotransplantation of connective tissue from a donor site to the site of recession.

SUMMARY:
This is an observational study. The participants in this study will be patients at the Graduate Periodontics Clinic at The Ohio State University who are planning to get a gingival graft to treat their gum recession. Gingival grafts are a common way to treat this recession. The grafting surgery is not part of the study.

The main purpose of this study is to better understand the normal healing of a gum graft. In order to do that, the investigators will take different kinds of measurements.

1. It is common for the tissue around the graft to have some swelling after the surgery. The investigators will measure the amount of swelling at different times as the graft heals. This will be done with a digital scanner which is passed over the area.
2. A device which measures blood flow will be used to see how new blood vessels are forming. This is also a device which is only passed over the area, so it is not invasive.
3. Saliva samples will be taken from around the teeth using sterile paper strips. This fluid will be analyzed for substances related to wound healing.
4. Participants will fill out questionnaires about their experience with the graft healing.

ELIGIBILITY:
Inclusion Criteria:

* Clinical (oral) Ohio State University College of Dentistry patient, treatment planned for SCTG procedure
* Miller Recession Class I, II, or III
* Teeth; Maxillary or mandibular incisors, canines, pre-molars
* Gingival Index ≤ 1
* Plaque Index ≤ 1
* Able and willing to provide informed consent
* Able and willing to complete questionnaire

Exclusion Criteria:

* Carious lesions on the tooth selected for surgical root coverage
* Taking any medications affecting the gingiva and/or oral mucosa: phenytoin, calcium channel blockers , cyclosporin A, immunostimulants/ immunomodulators
* Quantitative and/or qualitative defects on host inflammatory cells
* Organ transplant(s)
* Type I or II diabetes
* Currently pregnant or lactating
* Usage of smokeless tobacco
* Physical/mental handicap which can interfere with adequate oral hygiene performance

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The patients will be recruited from the patient pool of the Ohio State graduate periodontics clinic. These patients are referred to the Ohio State clinics to treat gum recession. Potential participants will be recruited after they have been treatment planned for subepithelial connective tissue grafting in the periodontics clinic. At the time of treatment planning, the investigators will present the option to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Tissue Volume Change | Immediately prior to surgery; immediately after surgery; Day 2 post-surgery; Day 3 post-surgery; Day 7 post-surgery; Day 14 post-surgery; Day 21 post-surgery
  3-dimensional digital scans will be taken with an intraoral scanner. Once captured, pre- and post-treatment digital image files will be overlapped and analyzed for dimensional changes in the area of the graft. Using digital software, the investigators will calculate the percentage tissue volume change between each time point, using the post-operative scan as a reference.
Correlation with Graft Exposure | Immediately prior to surgery; immediately after surgery; Day 2 post-surgery; Day 3 post-surgery; Day 7 post-surgery; Day 14 post-surgery; Day 21 post-surgery
  Surgical approaches for subepithelial connective tissue grafting can vary depending on site anatomical characteristics. The choice is often dictated by the anatomy of the site and the severity of the recession and sometimes by operator preference. For the purpose of this study, exposure of the graft will be analysed as an incidental occurrence as surgical needs dictate whether the graft will be exposed or not.
Inflammatory Cytokines | Immediately prior to surgery; immediately after surgery; Day 2 post-surgery; Day 3 post-surgery; Day 7 post-surgery; Day 14 post-surgery; Day 21 post-surgery
  Saliva samples will be taken from around the teeth at the surgical site by using sterile paper strips. These will be used to study the release of inflammatory cytokines.
Microvascular blood flow | Immediately prior to surgery; immediately after surgery; Day 2 post-surgery; Day 3 post-surgery; Day 7 post-surgery; Day 14 post-surgery; Day 21 post-surgery
  Laser Doppler Flowmetry (LDF) is a method of determining the real-time microvascular blood flow in soft tissue. LDF will allow the investigators to measure revascularization of the connective tissue graft and see if the degree of soft tissue dimensional change correlates with LDF measurements at certain time points.
Post-operative Pain and Analgesic Use | 2, 3, 7, 14 and 21 days after surgery
  A post-operative questionnaire will assess the subjects' post-operative pain using visual analog scales, including the location of the pain. The questionnaires will also assess the frequency and effectiveness of the analgesic prescribed.

SECONDARY OUTCOMES:
Thickness of the Gingival Flap and Graft | Day of surgery
  Gingival biotype refers to biological groupings of gingival phenotypes. Biotype has repeatedly been shown to influence clinical outcomes and tissue responses. In this study, the investigators will take biotype into account by measuring the thickness of the flap after it has been raised using tissue callipers. Additionally, the investigators will measure the thickness of the graft using the same method. These measurements will allow the investigators to determine if the biotype of the patient relates to the amount of edema post-surgery, and if that edema is primarily occurring in the flap or the graft itself.

CONTACTS AND LOCATIONS:
Overall Officials: Binnaz Leblebicioglu, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Graduate Periodontics Clinic, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No